CLINICAL TRIAL: NCT05681130
Title: Effect of Depression, Anxiety and Stress Scores on Embryo Transfer Success
Status: Completed | Type: Observational
Sponsor: Eurofertil IVF Health Center (Other)
Responsible Party: Sponsor
Other Study IDs: IVF- Stress
Record Dates: First submitted 2022-12-27; First posted 2023-01-12 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Stress; Pregnancy
Keywords: depression; anxiety; stress; pregnancy; IVF
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1 women attending IVF programme: Women attending to IVF programme will be evaluated for pscyhological parameters before and after the precedure
  Interventions: Other: questionaire
- 2 partners of women attending to IVF programme: Men who are partners of women attending to IVF programme will be evaluated for pscyhological parameters before and after the precedure
  Interventions: Other: questionaire

INTERVENTIONS:
Other: questionaire — two questionaires for each group

SUMMARY:
Psychological status of couples attending to IVF programmes is important due to possible effect on final result. Observers aim to investigate the depression, anxiety and stress scores of couples before and after the procedure.

DETAILED DESCRIPTION:
Studying effect of psychology on IVF is not a new idea. "Before and after" scores of women attending to IVF programmes had been studied numerous times. However, there is not sufficient data about the contbibution of male compartment upon the process. Investigators aimed to study both male and female participants. Final scores will not be evaluated unless at least good quality blastocsyt is transferred.

ELIGIBILITY:
Inclusion Criteria:

* 20 to 40 year old women attending to IVF programme

Exclusion Criteria:

* Azospermia and severe male factor for whom sperm freezing will be required
* History of RIF
* Known genetik abnormality of couples

Ages: 20 Years to 40 Years | Sex: All
Age Groups: Adult
Gender Based: Yes — reproductive aged women
Study Population: Women ages 20-40, without history of RIF or known genetic aneuploidy. Men without severe sperm problem without known genetic aneuploidiy. Only blastocyst transferred copules will be eligible for final analysis.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-02-17 (Actual); Study Completion 2024-02-17 (Actual)

PRIMARY OUTCOMES:
positive pregnancy test | 12 days after embryo transfer
  blood test will be taken after embryo (blastocyst) transfer

CONTACTS AND LOCATIONS:
Overall Officials: gerçek aydın, Study Director — Eurofertil IVF Health Center
Locations (1):
- Eurofertil, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
will be evaluated upon request